CLINICAL TRIAL: NCT06871735
Title: Acellular Collagen Matrix (Mucograft) as a Tool to Obtain Wound Closure Following GBR Procedures
Brief Title: Acellular Collagen Matrix as a Tool to Obtain Wound Closure Following a Guided Bone Regeneration Procedure
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Binnaz Leblebicioglu, Professor, Ohio State University
Other Study IDs: 2023H0107
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bone Graft
Keywords: GBR; Bone graft; dental implant
MeSH Terms: interventions — Wound Closure Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With acellular matrix: Participants who are having the GBR procedure done with the use of the acellular matrix material to cover the graft/wound
  Interventions: Procedure: Acellular matrix
- Surgical closure: Participants who are having the GBR procedure done by having the wound closed without the acellular material
  Interventions: Procedure: Surgical closure

INTERVENTIONS:
Procedure: Acellular matrix — Wound closure is obtained by use of acellular matrix material placed over the exposed barrier membrane. The procedure itself is not part of the research study, nor is the decision to use this procedure, but it is the condition of interest to the research.
  Groups: With acellular matrix
Procedure: Surgical closure — Wound from the graft is surgically closed, with no use of the acellular matrix. The procedure itself is not part of the research study, nor is the decision to use this procedure, but it is the condition of interest to the research.
  Groups: Surgical closure

SUMMARY:
Guided bone regeneration (GBR) is a procedure used to increase the amount of bone volume in the jaw before placing a dental implant. It is needed when a lot of bone has been lost around the spot where a tooth has been lost or extracted.

An incision is made, bone grafting material is placed in that spot, there is a membrane put over it as a barrier, then gum tissue has to be pulled back over it. Usually, this is enough to cover the whole wound, but sometimes the barrier membrane can't be covered with tissue the whole way without too much pulling, and the barrier membrane is still exposed.

In that case, one thing that can be done is to place another material, an acellular collagen matrix, over the barrier membrane and secure it there. This material has been shown to help with the healing in these cases.

Participants in this study will be clinic patients who have been determined to need a GBR procedure. Participants will get the GBR. If the barrier membrane is still exposed, then the acellular matrix material will be placed. This study will compare the healing outcomes and the success of the GBR depending on whether the acellular matrix material was used. The procedure itself is not part of the study. The only people in the study are patients who are already planning to have this procedure done as part of their dental care.

It is important to note that the research study will not affect the care that the patient is given, or whether or not the acellular matrix material is used. That will be decided by the dental surgeon who is treating them, based on their clinical judgement. The research study will only observe and compare the outcomes.

For the study, participants will have some additional clinical measurements made, besides the ones that are done as part of the follow-up care, and will be asked questions about their experience.

DETAILED DESCRIPTION:
Implant treatment planning is restorative driven. Thus, hard and soft tissue contours should be carefully studied based on ideal restorative treatment outcome. Any deficiency in supporting tissues has to be treated by using Guided Bone Regeneration (GBR) prior to implant placement. As defined in the Glossary of Periodontal Terms, GBR is a surgical procedure with the goal of augmenting bone volume in edentulous or peri-implant areas using a barrier membrane, often in conjunction with bone grafting materials and/or biologics. Wound closure following guided bone regeneration (GBR) procedure is essential to establish and maintain wound stability which is critical for targeted increase in bone volume. This can be accomplished, in general, by performing periosteal releasing with/without vertical incisions and by coronally positioning the flap. This manipulation, in turn, may create shallower vestibulum, less attached gingiva and muscle pull close to newly established alveolar crest.

Surgical site will be anesthetized with routine local anesthesia protocol. Crestal incisions followed by sulcular and/or vertical incisions will be performed, and full thickness flap elevation will be performed to reach alveolar bone. Recipient site will be prepared through decortication of the bone surface, trimming, and adapting the cross-linked collagen membrane. Allograft alone or mixed with autograft and/or xenograft will be placed into defect based on case specific indications. Wound closure will be accomplished by suturing the edges of the wound. In some cases, conventional method of wound closure through periosteal releasing incision and coronally positioned flap is not possible due to anatomical limitations. Although not ideal, barrier membrane is left exposed during healing for these cases. We intend to cover these exposed areas with ACM (acellular matrix) as described in the literature to determine whether this approach differentially affects outcomes. Standard post-operative care protocols will be followed including post-operative prescriptions for antibiotics, analgesics and antiseptic mouth rinse.

This clinical study aims to compare these two techniques by evaluating the clinical outcomes of early wound healing. The working hypothesis is that the use of acellular collagen matrix prevents shallow vestibulum formation and secondary surgeries to overcome with soft tissue deficiencies compared to conventional surgical approach.

Research related procedures: - Radiographic/CBCT and clinical measurements and recording of the alveolar ridge prior to surgery (these are obtained as part of standard of care to evaluate the site during treatment planning for bone grafting then, later, for implant placement. We will be recording additional volumetric measurements by using these tools [same radiographic/CBCT documents] as part of the study). - Clinical measurements and recording of the alveolar ridge dimensions after flap elevation and after ridge augmentation. - Details of the surgery including bone quality (reported by surgeon), presence of buccal dehiscence/fenestration, the need of additional bone grafting of the ridge, the indications for barrier membrane placement. - Soft and hard tissue sampling at implant placement surgery (these tissues are generally discarded while opening space for implant fixture. We intend to keep them to study the quality of the regenerated tissues). - Questions to evaluate patient experience (pain and discomfort during and after surgery).

Observation period will be up to 4-6 months (until implant placement surgery) and wound healing will be evaluated through clinical parameters (8-10 days, 6-8 weeks and 4-6 months), implant stability (initial and 4-6 months) and CBCT (pre-surgical and 4-6 months ridge dimensions). These post-operative observation periods are a part of standard protocol. Each appointment may be 40 minutes longer than routine appointment due to research related measurements.

ELIGIBILITY:
Inclusion Criteria:

* Have a missing tooth or teeth which are planned to be replaced with an implant
* Need for guided bone regeneration procedure to increase the bone available for implant placement
* Systemically healthy with no contraindications for bone grafting and/or implant surgery
* No chronic sinus problems
* Non-smoker
* No need for removable temporary restorations during wound healing.

Exclusion Criteria:

* Patients that have sufficient bone volume to perform implant placement through conventional drilling protocol without any pre-implant GBR procedure
* Indications for pre-implant/pre-GBR soft tissue grafting procedure to increase existing soft tissue contours
* The need to wear a removable temporary restoration during healing

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients at the Graduate Periodontics Clinic at The Ohio State University College of Dentistry who have been treatment-planned for a guided bone regeneration procedure prior to dental implant.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Healing Score Index 8-10 days | 8-10 days following the surgical procedure
  Healing Score Index (Pippi modification of Landry wound healing index):
  * presence/absence of redness;
  * presence/absence of granulation tissue;
  * presence/absence of suppuration;
  * presence/absence of swelling;
  * degree of tissue epithelialization (partial/complete);
  * presence/absence of bleeding;
  * presence/absence of pain on palpation.
  * presence/absence of plaque (% of plaque positive surfaces)
  At first PO appointment
Healing Score Index 6-8 weeks | 6-8 weeks following the surgical procedure
  Healing Score Index (Pippi modification of Landry wound healing index):
  * presence/absence of redness;
  * presence/absence of granulation tissue;
  * presence/absence of suppuration;
  * presence/absence of swelling;
  * degree of tissue epithelialization (partial/complete);
  * presence/absence of bleeding;
  * presence/absence of pain on palpation.
  * presence/absence of plaque (% of plaque positive surfaces)
  At second PO appointment
Wound Healing 8-10 days | 8-10 days following the surgical procedure
  Clinical wound healing will be scored as yes or no for each of the following wound healing parameters:
  * Mature wound healing, defined as complete wound closure without other significant findings.
  * Erythema, defined as increased redness compared to adjacent non-operated sites
  * Bleeding, defined as presence of spontaneous bleeding at the wound site
  * Graft mobility, defined as loose subgingival bone graft material evaluated by gentle palpation using a UNC-15 probe (if grafting was done during surgery)
  * Suppuration, defined as presence of pus or discharge at the wound site
  * Necrosis, defined as any visual soft and/or hard tissue necrosis at the wound site
  * Clinical wound exposure and closure and hydrogen peroxide test(+/-)
  At first PO appointment
Wound Healing 6-8 weeks | 6-8 weeks following the surgical procedure
  Clinical wound healing will be scored as yes or no for each of the following wound healing parameters:
  * Mature wound healing, defined as complete wound closure without other significant findings.
  * Erythema, defined as increased redness compared to adjacent non-operated sites
  * Bleeding, defined as presence of spontaneous bleeding at the wound site
  * Graft mobility, defined as loose subgingival bone graft material evaluated by gentle palpation using a UNC-15 probe (if grafting was done during surgery)
  * Suppuration, defined as presence of pus or discharge at the wound site
  * Necrosis, defined as any visual soft and/or hard tissue necrosis at the wound site
  * Clinical wound exposure and closure and hydrogen peroxide test(+/-)
  At second PO appointment

SECONDARY OUTCOMES:
Change in ridge dimension | Day of surgery, 1st PO appt (8-10 days post surgery), 2nd PO appointment (6-8 weeks post surgery), final appointment (4-6 months post surgery)
  Ridge height and width, measured using the surgical template
Patient experience - surgery | Day of surgical procedure
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain) Any postsurgical issues reported
Patient experience - 8-10 days PO | 8-10 days following the surgical procedure
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any postsurgical issues reported
  At first post-op appointment
Patient experience - 6-8 weeks PO | 6-8 weeks following the surgical procedure
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any postsurgical issues reported
  At second post-op appointment
Patient experience - implant appointment | 4-6 months following the surgical procedure
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any postsurgical issues reported
  At second post-op appointment

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Graduate Periodontics Clinic, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No